CLINICAL TRIAL: NCT07130747
Title: Effect of Myofascial Release Versus Deep Friction Massage on Abdominal Recovery and Scar After Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moaz khaled elsayed mohamed rousha, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moaz_Msc
Record Dates: First submitted 2025-08-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myofascial Release; Deep Friction Massage; Cesarean Section Complications; Scar
MeSH Terms: conditions — Cicatrix | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home advices (Active Comparator): It consisted of 12 postpartum women having a post-Cesarean-section scar. They will receive no treatment program, only advices for home care
  Interventions: Other: Routine daily scar care advices
- myofascial release technique (Experimental): It consisted of 12 postpartum women having a post-Cesarean-section scar. They will receive myofascial release technique for 20 minutes three times per week for eight weeks, in addition to advices for home care
  Interventions: Other: Myofascial release; Other: Routine daily scar care advices
- deep friction massage (Experimental): It consisted of 12 postpartum women having a post-Cesarean-section scar. They will receive deep friction massage for 20 minutes three times per week for eight weeks, in addition to advices for home care.
  Interventions: Other: Deep friction massage; Other: Routine daily scar care advices

INTERVENTIONS:
Other: Myofascial release — The study involves women in both groups receiving myofascial release technique for twenty minutes three times per week for eight weeks. The technique requires the patient's skin to be dry and not oily, and all techniques must be applied at the barrier of tissue resistance. The technique involves gentle, sustained pressure held at the barrier for at least five minutes to allow the patient to respond to the treatment and relax. The technique involves skin stretching and desensitization around the scar, using up and down, side-to-side, and circular maneuvers.
  Arms: myofascial release technique
Other: Deep friction massage — Women in both groups (C) will receive a deep friction massage three times a week for eight weeks, applying a fingertip pad perpendicularly to post-cesarean scar tissue, moving across the band and back-and-forth motion along the scar tissue's length.
  Arms: deep friction massage
Other: Routine daily scar care advices — Each woman in all groups (A, B, and C) will receive full instructions for daily post-cesarean-section scar care. Weekly revision for post-cesarean-section scar care will conduct by the researcher

SUMMARY:
This study was done to compare the effect of myofascial release versus deep friction massage on abdominal recovery and scar after cesarean section.

DETAILED DESCRIPTION:
Chronic post-C-section scar pain and discomfort affect up to 20% of women who undergo cesarean sections. This pain can lead to physical, aesthetic, psychological, and social consequences, including itching, stiffness, scar contractures, and tenderness. The myofascial release technique, a manual approach, may facilitate the healing process. Deep friction massage, used to correct structural alterations, can cause reduced mobility and viscoelasticity, potentially affecting sensory receptors and nerve fibers. This study aims to provide physiotherapists with scientific information on the effect of myofascial release on scar and abdominal recovery after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

1. All postpartum women >6 months postnatal having a post-Cesarean-section scar.
2. Postpartum women with a well-healed cesarean section scar resulted in chronic pain in the scar, pelvis, or abdomen.
3. Their ages will range from 30 to 45 years.
4. Their body mass index (BMI) is less than 30 kg/m².

Exclusion Criteria:

1. Pregnant women or planning for pregnancy.
2. Postpartum women with abdominal infectious diseases.
3. Cardiovascular diseases.
4. Previous spinal surgery.
5. History of skeletal deformity.
6. Participation in any other exercise training program during this study.
7. Malignant condition
8. History of acute infection
9. Neurological problem
10. Mental problem to prevent evaluation and cooperation
11. Having uncontrolled metabolic diseases like diabetes and thyroid disease

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All postpartum women >6 months postnatal having a post-cesarean-section scar. Their ages will range from 30 to 45 years
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
assessment of pain intensity | at baseline and after 8 weeks
  Participants will use a visual analogue scale to assess waist pain intensity before and after treatment for all groups, rating severity from zero to 10. This reliable and time-efficient method is suitable for assessing pain levels post-c Cesarean scar site.

SECONDARY OUTCOMES:
Assessment of post-Cesarean-section scar recovery | at baseline and after 8 weeks
  The modified Vancouver scale will be used to assess post-Cesarean section scar tissue, focusing on vascularity, pigmentation, pliability, and height. The scale will be tested using four characteristics of the scar: vascularity, height, pliability, and pigmentation. The overall score between 0 and 13 is calculated by adding up the scores of each characteristic. The modified scale will be evaluated through multiple photographs of the patient's scar, evaluating four parameters: irregularity of texture, height, pigmentation, and vascularity. Modifications may be suggested to improve reliability and teaching, but it is not yet a validated tool.
Assessment of pressure pain threshold | at baseline and after 8 weeks
  A pressure algometer is a reliable device used to assess pressure pain threshold and deep tenderness in post-Cesarean scar tissue. It consists of a gauge attached to a rubber tip and calibrated in kg/cm², with a range of 1-10 kg/cm². The algometer has a probe, handheld and analogue pieces, and measures accurately to 0.1 kg/cm². Participants are instructed to relax in a comfortable supine position, and the pressure is increased by one kilogram per second until discomfort is felt. The mean pressure value is recorded as the pressure pain threshold at the post-Cesarean scar.
Assessment of abdominal recovery | at baseline and after 8 weeks
  The study will conduct an abdominal endurance test for all participants pre- and post-treatment. Participants will lie with a 70° wooden support, and the researcher will measure their endurance and functional ability. If they cannot sustain their position, they will be recorded as having poor endurance and functional ability, while those who can sustain their position for 15-30 seconds will be classified as having perfect endurance and functional ability.
Assessment of abdominal musculatures strength | at baseline and after 8 weeks
  The study will conduct a manual muscle test on all participants pre- and post-treatment, assessing abdominal musculature strength using Dr. Lovett's manual muscle test scale. The rectus abdominus muscle will be examined by lifting the participant to the lower end of the scapulae, leaning forward with crossed hands, and repeating this motion. The test will be recorded on a 0-5-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- the Gynecology and Obstetrics Outpatient clinics, Alexandria University Hospitals, Alexandria, Egypt, Alexandria, Egypt